CLINICAL TRIAL: NCT03070561
Title: Evaluating the Placement of a Peanut Immunotherapy Dissolving Film in Healthy Subjects
Brief Title: Evaluating Peanut Immunotherapy Dissolving Film in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JHU NA_00072576
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Peanut Allergy; Immunotherapy; Pharmacokinetics
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Open label, crossover, local pharmacokinetics study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sublingual film with peanut extract (Experimental)
  Interventions: Biological: sublingual film with peanut extract

INTERVENTIONS:
Biological: sublingual film with peanut extract

SUMMARY:
Open label, cross-over, local pharmacokinetics study of a sublingual film with peanut extract in healthy adults and children

DETAILED DESCRIPTION:
In this study, 15 non-peanut allergic children and adults will be enrolled. At three visits, each at least a day apart, the study product (dissolving film) containing approximately 60 mcg of the major peanut allergen (Ara h 2), equivalent to approximately 1000 mcg of peanut protein, will be placed in one of three areas: the sublingual space, affixed to the buccal mucosa, and in the vestibular space. Concentrations of Ara h2 in saliva collected at several locations over several time points in the mouth will be analyzed by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years and <30 years.
* Able to give informed consent.
* English speaking with no language impairment
* Regularly consume a meal sized portion (approximately 5 grams) of peanut at least twice per month during the preceding 6 months

Exclusion Criteria:

* History of reaction to peanuts
* Major active medical problems of the oral cavity or use of medications that might change rates of salivation

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Measurement of elimination half life (T1/2) of the Ara H2 in sublingual placement | 3 days
Measurement of elimination half life (T1/2) of the Ara H2 in buccal placement | 3 days
Measurement of elimination half life (T1/2) of the Ara H2 in vestibular placement | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Keet, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No